CLINICAL TRIAL: NCT04864665
Title: A Prospective, Multicentre Before and After Study to Evaluate the Effects of a Formula With Prebiotics and Milk Fat, on the Gut Health of Chinese Infants and Young Children
Brief Title: Study to Evaluate the Effects of a Formula on the Gut Health of Healthy Chinese Infants and Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Collaborators: Nutricia Early Life Nutrition (Shanghai) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SBB0E_34098
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Healthy Children
Keywords: Prebiotics; Gut microbiota; Formula
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: interventional with breastfed reference group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formula fed (Experimental): 0 - 6 months: a formula with prebiotics and milk fat (Stage 1); >6 - 12 months: a formula with prebiotics and milk fat (Stage 2); >1 - 2 years: a formula with prebiotics and milk fat (Stage 3)
  Interventions: Dietary Supplement: a formula with prebiotics and milk fat

INTERVENTIONS:
Dietary Supplement: a formula with prebiotics and milk fat — Provided in a formula added with prebiotics and milk fat for 1 month

SUMMARY:
The infant gut microbiota, a major driver of the maturation of the immune system, is formed through the successive establishment and development during infancy and early childhood. It can inhibit the growth of pathogenic bacteria, prevent the occurrence of diseases and improve the child's quality of life. It is therefore important to regulate the microbiota balance in infants and young children.

This objective of this post-launch study is to evaluate the effects of a formula with prebiotics and milk fat on the gut microbiota and stool characteristics of healthy Chinese infants and young children. The duration of the study for each participant is 32 days and includes 3 study visits.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age was 37-42 weeks at birth;
* Birth weight ≥2,500 g and ≤ 4,500 g;
* Chinese nationality;
* Weight and height are within normal range (i.e. WHO Child Growth Standards

  * 2SD);
* No relocation across provinces/ cities in the past 1 year and no plans to relocate during the study period.
* Breastfeeding reference: breastfeeding at the time of enrollment, and the mother intends to continue breastfeeding throughout the study period;
* Intervention arm: formula feeding / habitual milk drinking (formula milk, milk and other dairy products) at the time of enrollment, and willing to change from the original milk powder / dairy product to the study formula, and consume it as instructed during the study period;
* The child's parent(s) / guardian has access to a mobile phone on which the secure digital WeChat platform can be installed and used, connect to the network, take photographs and record defecation, and complete questionnaires during the study;
* The child's parent(s) / guardian is of legal age of consent, has sufficient command of Chinese (Mandarin) language to complete the informed consent and other study documents, is willing and able to fulfill the requirements of the study.
* The child's parent(s) / guardians can be contacted directly by telephone or WeChat;

Exclusion Criteria:

* Neonatal asphyxia at birth;
* Chronic infectious, metabolic, genetic illness or other disease including any condition that impacts feeding or may impact study outcomes;
* Cognitive and developmental disorders;
* Antibiotic usage up to 2 weeks before enrollment;
* Ongoing antibiotic treatment;
* Taking probiotic supplements or formula with probiotics up to 1 month before enrollment;
* Participation in other clinical trials;
* Parent(s)' / guardian's refusal to participate in the study;
* Known or suspected allergy to cow milk, soy or fish

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 455 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Change in stool bifidobacteria level | 32 days
  Stool sample analysis

SECONDARY OUTCOMES:
Change in stool lactobacillus level | 32 days
  Stool sample analysis
Change in stool characteristics | 32 days
  • Stool image analysis based on the 4-point Brussels Infant and Toddler Stool Scale (watery, loose, formed, hard, with hard stools indicating worse outcome)
Change in gastrointestinal tolerance | 32 days
  Parent reported questionnaire
Satisfaction with the study product | 32 days
  Parent reported questionnaire

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Zhengzhou Children's hospital of Henan Children's hospital, Zhengzhou, Henan
  - Tangdu Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang
  - Beijing Children's Hospital of Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No